CLINICAL TRIAL: NCT01698346
Title: Impact of Pertussis Vaccination in Pregnancy on Maternal Protection Offered to Young Infants
Brief Title: Pertussis (Tdap) Vaccination in Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Responsible Party: Principal Investigator, Elke Leuridan, MD, PhD, MD, PhD, Universiteit Antwerpen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: cev001; 2011-001936-45 (EudraCT Number)
Record Dates: First submitted 2012-09-21; First posted 2012-10-03 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Pertussis; Pregnancy
Keywords: Pertussis; Infants; Vaccination; Pregnancy
MeSH Terms: conditions — Whooping Cough | interventions — Pertussis Vaccine; Boostrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): 50 unvaccinated pregnant women
- Pertussis vaccine (Boostrix®, GSK Biologicals, Rixensart) (Active Comparator): 50 pregnant women vaccinated with pertussis vaccine
  Interventions: Biological: Pertussis vaccine

INTERVENTIONS:
Biological: Pertussis vaccine — Vaccination during pregnancy with a pertussis containing vaccine
  Other Names: Boostrix®, GSK Biologicals, Rixensart
  Arms: Pertussis vaccine (Boostrix®, GSK Biologicals, Rixensart)

SUMMARY:
Despite good vaccination coverage, included in national immunization programs in developed countries, the number of reported pertussis cases is rising, also in very young infants. Current immunization strategies fail to protect infants too young to be immunized with the licensed vaccine. Different strategies are possible to close the gap of susceptibility between the loss of maternal antibodies and protection by vaccination. The main aim of the present study is to measure the influence of an adult pertussis booster in pregnant women, on the titer and duration of maternal antibodies in their infants. Early humoral immunity will be assessed and the influence on vaccine response of the infant measured. The present study offers the opportunity to have new insights in neonatal immunological mechanisms against pertussis and a better understanding in strategies to protect infants against pertussis.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-35 years
* Willing to be immunized during pregnancy OR
* Received already a pertussis vaccination during pregnancy, as advised by gynaecologist or general practitioner.
* Age matched controls will be identified in the same time period in the recruiting hospital.
* Availability for follow-up visits and phone call access through 16 months following delivery
* Willing to have infant immunized with hexavalent vaccine at 8.12 and 16 weeks and 15 months of age (= normal Belgian schedule) with pediatrician, the general practitioner or at the Centre for the Evaluation of Vaccination.
* In the 18th-32nd week of a pregnancy at low risk for complications as determined by the obstetrician

Exclusion Criteria:Women:

* Serious underlying medical condition
* History of a febrile illness (>= 38° Celsius) within the past 72 hours before injection
* Previous severe reaction to any vaccine
* Receipt of tetanus-diphtheria toxoid immunization within the past 1 month
* Receipt of tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine absorbed (Tdap) immunization in the last 10 years
* Receipt of a vaccine, blood product (excluding Rhogam) or experimental medicine within the 4 weeks prior to injection through 4 weeks following injection
* Receipt of or plans to receive influenza vaccine within the 4weeks prior to or following injection. One month interval should be respected in order to evaluate eventual Adverse events following one of both vaccines (fever, local symptoms).
* High risk for serious obstetrical complication
* Anything in the opinion of the investigator that would put the participant at risk.

Exclusion criteria for the offspring:

* Serious underlying medical condition
* No signed informed consent by both parents
* Severe reactions to any vaccine
* Anything in the opinion of the investigator that would put the participant at risk.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2012-02; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Does vaccination of pregnant women with a combined vaccine Tetanus, diphtheria and acellular pertussis (Tdap), induce sufficiently high maternal antibody concentration in the newborns infants to possibly protect them until their own vaccination starts | 16 months
  1. What are the concentrations of IgG against Pertussis Toxin (anti-PT), Filamentous Haemagglutinin (anti-FHA), Fimbriae (anti-Fim) and pertactin (anti-PRN):
     1. in women during pregnancy and at delivery after vaccination with TdaP
     2. in children at birth (cord), before starting vaccination (week 8), one month after primary course of three doses (week 20) and before and after the fourth pertussis vaccine dose (at month 15 and 16)
  2. What are the concentrations of anti-tetanus and anti-diphtheria IgG antibodies at all mentioned time points, to evaluate interference when administering several antigens and to evaluate the influence of maternal antibodies on vaccine response to tetanus and diphtheria in infants

SECONDARY OUTCOMES:
Vaccine associated (Severe) Adverse Events ((S)AE) in pregnant women and children during the study time | 16 months
  Vaccine associated (Severe) Adverse Events ((S)AE) in pregnant women and children during the study time
Infant growth measurement at all time points | 16 months
  Infant growth measurement at all time points
Assessment of pneumococcal immune response in infants whose mothers received Tdap vaccination during pregnancy | 12 months
  The present trial on pertussis vaccination during pregnancy, offers the opportunity to add evidence for a possible blunting effect of infant immune responses to pneumococcal infant vaccination after maternal Tdap vaccination. Pneumococcal antibodies will be measured in serum samples taken from infants after a primary series of 2 pneumococcal vaccine doses (2 and 4 months of age) and after a third vaccine dose (at 12 months of age). Infants are born from either vaccinated or unvaccinated mothers.

CONTACTS AND LOCATIONS:
Overall Officials: Elke Leuridan, MD, PhD, Principal Investigator — Universiteit Antwerpen; Thu Ha Thi Hoang, MD PhD, Principal Investigator — National Institute for Hygiene and Epidemiology
Locations (2):
- Centre for the Evaluation of Vaccination, Antwerp, Belgium
- National Institute of Hygien and Epidemiology, Hanoi, Vietnam

REFERENCES:
- [Derived] Maertens K, Cabore RN, Huygen K, Vermeiren S, Hens N, Van Damme P, Leuridan E. Pertussis vaccination during pregnancy in Belgium: Follow-up of infants until 1 month after the fourth infant pertussis vaccination at 15 months of age. Vaccine. 2016 Jun 30;34(31):3613-9. doi: 10.1016/j.vaccine.2016.04.066. Epub 2016 Apr 30. PMID 27142328